CLINICAL TRIAL: NCT04819945
Title: A Prospective, Multicenter, Single-arm, Clinical Investigation Evaluating the Safety and Performance of GATT-Patch for Hemostasis During Open Liver Surgery
Brief Title: Clinical Safety and Performance of GATT-Patch in Open Liver Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GATT Technologies BV (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF-01-QR-021
Record Dates: First submitted 2021-03-17; First posted 2021-03-29 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Hemorrhage, Surgical
Keywords: Hemostatic patch; Surgical sealant; Open Liver Surgery; Hemostasis
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GATT-Patch (Experimental): GATT-Patch will be used to control bleeding during open liver surgery. Each surgery will be performed according to the standard procedures at the hospital, with the exception of the use of GATT-Patch.
  Interventions: Device: GATT-Patch

INTERVENTIONS:
Device: GATT-Patch — Use of GATT-Patch for minimal, mild or moderate bleeding sites in open liver surgery

SUMMARY:
The purpose of this study is to determine the clinical safety and performance of GATT-Patch for management of haemorrhage during elective open liver surgery.

DETAILED DESCRIPTION:
The GATT-Patch study is a prospective, single arm, multicenter, pre-market, first-in-man clinical investigation, that intents to determine the clinical safety and performance of GATT-Patch for management of haemorrhage during elective open liver surgery.

The clinical investigation will be carried out in a maximum of 7 sites in The Netherlands, treating an estimated total of 51 participants. All participants will be thoroughly screened and if found eligible, treated with GATT-Patch during open liver surgery. Participants will be followed for 6 weeks with an additional ultrasound assessment at the 6 week follow up visit.

The participant enrolment period is expected to take approximately 6 months, with a total expected duration of the clinical investigation of approximately 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant is scheduled to undergo an elective open surgery on the liver;
* Participant is willing and able to give written informed consent for investigation participation;
* Participant is 18 years of age or older at the time of enrollment;
* Participant has been informed of the nature of the clinical investigation.

A participant must meet all of the following intraoperative inclusion criteria to be treated with the investigational device:

* Participant in whom the Investigator is able to identify a target bleeding site at the liver resection plane for which any applicable conventional means for hemostasis (e.g. suture, ligature or cautery) are ineffective or impractical and the choice is made to use a topical hemostat for control of hemostasis; and the choice is made to use a topical hemostat for control of hemostasis;
* Participant has a minimal, mild, or moderate target bleeding;

Exclusion Criteria:

* Participant is scheduled to undergo surgery on other organs besides the liver (e.g. pancreas, colon, lungs);
* Participant is taking multiple antithrombotic therapies in therapeutic dosage up to the time of surgery, allowing exclusive use of acetylsalicylic acid;
* Participant has platelet count <100 x 10ˆ9/L, an activates partial thrombin time of >100s, or international normalized ratio >2.5;
* Participant is pregnant, planning on becoming pregnant or actively breast-feeding during the follow-up period;
* Participant has a known hypersensitivity to brilliant blue (FD&C Blue #1);
* Participant has an active or suspected infection at the surgical site;
* Participant has a total bilirubin level of ≥ 2.5 mg/dl
* Participant has had or has planned to receive any organ transplantation;
* Participant has American Association of Anesthesiologists (ASA) classification of 4/5;
* Participant has a life expectancy of less than 3 months;
* Participant has a documented severe congenital or acquired immunodeficiency;
* Participant in whom the investigational device will be used at the site of a synthetic graft or patch implant;
* Participant is currently participating or has participated in another clinical investigation within the past 30 days that may affect the endpoints of the study, such as trials related to the surgical procedure, and on anti-coagulation;
* Participant is not appropriate for inclusion in the clinical investigation, per the medical opinion of the Investigator;
* Participant has any incidental (pre- and peri-operative) findings deemed by the Investigator to potentially jeopardize the safety or welfare of the patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Head, MD PhD, Study Director — GATT Technologies BV; Hans de Wilt, Prof. dr., Principal Investigator — Radboud University Medical Center; Harry van Goor, Prof. dr., Study Chair — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Erasmus University Medical Center, Rotterdam, South Holland
  - University Medical Center Groningen, Groningen

REFERENCES:
- [Derived] de Wilt JHW, Verhoef C, de Boer MT, Stommel MWJ, van der Plas-Kemper L, Garms LM, van der Zijden CJ, Head SJ, Bender JCME, van Goor H, Porte RJ. Clinical Safety and Performance of GATT-Patch for Hemostasis in Minimal to Moderate Bleeding During Open Liver Surgery. J Surg Res. 2024 Jun;298:316-324. doi: 10.1016/j.jss.2024.03.033. Epub 2024 Apr 18. PMID 38640617
- [Derived] Roozen EA, Lomme RMLM, Calon NUB, Ten Broek RPG, van Goor H. Efficacy of a novel polyoxazoline-based hemostatic patch in liver and spleen surgery. World J Emerg Surg. 2023 Mar 14;18(1):19. doi: 10.1186/s13017-023-00483-x. PMID 36918896

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 56 patients provided informed consent. There were 47 patients that received GATT-Patch during surgery.
Groups:
- GATT-Patch: GATT-Patch will be used during Stage I of the trial, after which a pause of the trial will take place for an independent safety assessment by the Data Monitoring Committee. If approved, GATT-Patch will furthermore be used during Stage II of the trial, which will include 39 patients for the primary endpoint analysis of hemostasis.
Period: Overall Study
Arm/Group | GATT-Patch
Started | 47
Completed | 46
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | GATT-Patch
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 43
  More than one race | 0
  Unknown or Not Reported | 2
Previous abdominal surgery, % [Count of Participants; unit: Participants] | 29
Hereditary blood disorders, % [Count of Participants; unit: Participants] | 1
Hemoglobin, g/dL [Mean (Standard Deviation); unit: g/dL] | 8.3 (0.8)
Platelet count, 10^9/L [Mean (Standard Deviation); unit: 10^9 platelets/L] | 219.4 (79.1)
Total bilirubin, umol/L [Mean (Standard Deviation); unit: umol/L] | 9.3 (4.9)
Indication for surgery [Count of Participants; unit: Participants]
  Colorectal carcinoma metastases | 31
  Hepatocellular carcinoma | 5
  Cholangiocarcinoma | 4
  Non-colorectal carcinoma metastases | 4
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Hemostasis
Description: Performance of GATT-Patch in achieving hemostasis at 3 minutes
Time Frame: During procedure
Measure: Count of Participants; unit: Participants
Groups:
- GATT-Patch Stage II Patients: Stage II of the trial was used for the primary endpoint analysis of hemostasis, and included 39 patients.
- GATT-Patch All Patients: All 47 patients treated with GATT-Patch during Stage I and Stage II of the trial.
Arm/Group | GATT-Patch Stage II Patients | GATT-Patch All Patients
Number analyzed (Participants) | 39 | 47
Participants | 38 | 46

2. Secondary Outcome: Mean Time to Hemostasis (Seconds)
Description: The mean time to hemostasis will be calculated based on time to hemostasis determined at 30 seconds intervals.
Time Frame: During procedure
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | GATT-Patch
Number analyzed (Participants) | 39
seconds | 54.6 (107.5)

3. Secondary Outcome: Hemostasis at Different Timepoints
Description: The number of participants achieving hemostasis at 30, 60, 90, 120, and 150 seconds will be determined.
Time Frame: During procedure
Measure: Number; unit: participants
Arm/Group | GATT-Patch Stage II Patients
Number analyzed (Participants) | 39
participants
  Hemostasis at 30 seconds | 32
  Hemostasis at 1 minute | 37
  Hemostasis at 90 seconds | 37
  Hemostasis at 120 seconds | 37
  Hemostasis at 150 seconds | 37
  Hemostasis at 3 minutes | 38

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to a 6-week (+ / - 2 weeks) follow-up visit.
Description: All events occurring during hospitalization after surgery, as well as occurring within the follow-up timeframe up to the 6-week follow-up visit were marked as adverse events. During hospitalization, systematic physical exams and laboratory assessments were performed and at 6 weeks an abdominal ultrasound was performed.
Arm/Group | GATT-Patch All Patients
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 7/47
Other Adverse Events (participants affected / at risk) | 14/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GATT-Patch All Patients (N=47)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Biloma (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Bile leakage (Hepatobiliary disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GATT-Patch All Patients (N=47)
Biloma / bile leakage (Hepatobiliary disorders) | 10 (10)
Hepatic hematoma (Injury, poisoning and procedural complications) | 4 (4)

LIMITATIONS AND CAVEATS:
This was a single-arm trial comparing GATT-Patch to a literature-derived performance goal. A randomized controlled trial will provide further insights into the performance of GATT-Patch versus a standard of care hemostatic patch.

The trial was performed at 3 sites and results may have been dependent on the experience of surgeons in using hemostatic agents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/45/NCT04819945/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT04819945/SAP_001.pdf